CLINICAL TRIAL: NCT06731829
Title: A Multicenter, Randomized, Double-Blind, Positive-Controlled, Cross-Over, Dose-Escalation Phase II Clinical Trial Evaluating the Efficacy and Safety of HRS-9231 for Central Nervous System (CNS) Magnetic Resonance Imaging (MRI)
Brief Title: A Study for Adults Undergoing Magnetic Resonance Imaging (MRI) for Known or Highly Suspected Brain and/or Spinal Cord Conditions
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: HRS-9231-201
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: For Contrast-enhanced Magnetic Resonance Imaging (MRI) of Central Nervous System (CNS) Lesions
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-9231 dose 1 (Experimental)
  Interventions: Drug: HRS-9231
- HRS-9231 dose 2 (Experimental)
  Interventions: Drug: HRS-9231
- HRS-9231 dose 3 (Experimental)
  Interventions: Drug: HRS-9231
- Gadobutrol (Active Comparator)
  Interventions: Drug: Gadobutrol

INTERVENTIONS:
Drug: HRS-9231 — HRS-9231
  Arms: HRS-9231 dose 1; HRS-9231 dose 2; HRS-9231 dose 3
Drug: Gadobutrol — Gadobutrol
  Arms: Gadobutrol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HRS-9231 for Central Nervous System (CNS) Magnetic Resonance Imaging (MRI); to explore the effective dose of HRS-9231 for CNS MRI; and to explore the population pharmacokinetic characteristics of HRS-9231 in CNS MRI subjects

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form, willing to cooperate with the study, and comply with trial requirements
2. Age ≥18 years, no gender restrictions
3. Known or highly suspected CNS lesions, with imaging showing at least one enhanced lesion
4. Scheduled for CNS contrast-enhanced MRI for clinical needs and agree to complete two contrast-enhanced MRI scans

Exclusion Criteria:

1. Clinically unstable condition or severe diseases that may affect trial results, such as inability to ensure imaging comparability or reliability of study parameters
2. Moderate to severe renal dysfunction, defined as aGFR < 60 mL/min
3. Contraindications to MRI, such as metallic implants or claustrophobia
4. History of severe allergies, including drugs, contrast agents, or other allergens
5. Severe liver disease or cardiovascular disease, or related abnormal test results
6. Central nervous system inflammation or recent history of stroke
7. Active infectious diseases, such as HIV, hepatitis B, or syphilis
8. Use of other contrast agents before or after study drug administration, or recent interventional treatments that may affect imaging comparability
9. Pregnancy, breastfeeding, or plans for conception, without effective contraception measures
10. Recent participation in other clinical trials or previous participation in studies involving gadolinium-based contrast agents
11. Other conditions deemed unsuitable by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Calculate the Contrast-to-Noise Ratio (CNR) based on the Signal Intensity (SI) of CNS lesions in MRI images after receiving HRS-9231 or the control drug (Gadobutrol) | 1 day procedure

SECONDARY OUTCOMES:
Medical applicability of MRI imaging for CNS lesions after receiving HRS-9231 or the control drug (Gadobutrol). | 1 day procedure
Number, size, and location of CNS lesions in MRI images after receiving HRS-9231 or the control drug. | 1 day procedure
Visualization scores for CNS lesions in MRI images after receiving HRS-9231 or the control drug (Gadobutrol): boundary delineation, internal morphology, and contrast enhancement. | 1 day procedure
HRS-9231 plasma concentration and population pharmacokinetic parameters (such as clearance, apparent volume of distribution, etc.). | 1 day procedure

CONTACTS AND LOCATIONS:
Locations (1):
- People's Hospital, Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided